CLINICAL TRIAL: NCT04242121
Title: The Risk Stratification in Patients With Multiple Myeloma Based on Fluorescence Flow Cytometry Quantitative Determination of the Circulating Plasma Cells in the Peripheral Blood
Status: Terminated | Type: Observational
Why Stopped: poor recruitment
Sponsor: Ivan S Moiseev (Other)
Responsible Party: Sponsor-Investigator, Ivan S Moiseev, Vice-director for science R.M. Gorbacheva Memorial Institute for Pediatric Oncology, Hematology and Transplantation, St. Petersburg State Pavlov Medical University
Organization: St. Petersburg State Pavlov Medical University (Other)
Other Study IDs: 222/2019
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Myeloma Multiple
MeSH Terms: conditions — Multiple Myeloma | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: fluorescence flow cytometry — Countification of plasma cells by fluorescence flow cytometry (hematology analyzer XN-1000/20)

SUMMARY:
The main aim of this study is to evaluate the effectiveness of the clinical application of the XN-1000/20 hematology analyzer for risk stratification in patients with multiple myeloma based on the number of detected plasma cells in peripheral blood at the different stages of treatment. This clinical study is observational and does not involve drugs. 100 subjects with newly diagnosed multiple myeloma will be enrolled in this study and followed for 3 years.

DETAILED DESCRIPTION:
The presence of circulating plasma cells in patients with multiple myeloma is considered as a marker for highly proliferative disease and associated with a worse prognosis.

Plasma cell counting is conventionally done by means of peripheral blood film morphology using light microscopy. However, this manual method is laborious as well as imprecise due to the low number of cells counted, and inter-observer variability. Flow cytometry with monoclonal antibodies is unsuitable as a screening test. The procedure is not automated, and it is expensive and time consuming. Therefore, new rapid, effective and inexepensive methods are needed for risk-stratification in patients with multiple myeloma.

Automated antibody-synthesizing or secreting cells counting from routine haematology systems (XN-1000/20) without sample preparation and in less than 1 minute will further reduce the workload in haematology laboratories and it can be used for counting circulating plasma cells in peripheral blood in patients with multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Newly diagnosed symptomatic multiple myeloma
* Signed informed consent
* No second tumors

Exclusion Criteria:

* Monoclonal gammopathies of undefined significance
* Smoldering Multiple Myeloma
* Plasma cell leukemia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed multiple myeloma (both with and withous auto-SCT groups) at the different stages of treatment
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Time-to-progression according to circulating plasma cells | [Time Frame: 3 years]
  Measured by cumulative incidence estimates

SECONDARY OUTCOMES:
Progression-free survival | [Time Frame: 3 years]
  Measured by Kaplan-Meier estimates
Overall survival | [Time Frame: 3 years]
  Measured by Kaplan-Meier estimates

CONTACTS AND LOCATIONS:
Locations (1):
- Boris V Afanasyev, MD, Prof., Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No